CLINICAL TRIAL: NCT00052195
Title: DARDAR Health Project (Disseminated Tuberculosis and HIV Infection)
Brief Title: Investigational Vaccine for the Prevention of Disseminated Tuberculosis in HIV Infected People
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, C. Fordham von Reyn, Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1R01AI045407-01A2 (NIH); 1R01AI045407-01A2 (NIH); 3R01AI045407-02S1 (NIH); 5R01AI045407-03 (NIH); U01AI045407-06 (NIH); U01AI045407-07 (NIH); U01AI045407-08 (NIH)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Tuberculosis; HIV Infections
Keywords: Mycobacterium vaccae; BCG; Disseminated tuberculosis; SRL-172; DAR-901
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — SRL172

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Placebo Comparator)
  Interventions: Biological: SRL-172
- A (Experimental)
  Interventions: Biological: SRL-172

INTERVENTIONS:
Biological: SRL-172 — 5 doses of 0.1mL vaccine or placebo given intradermally over 12-months

SUMMARY:
A significant number of HIV infected patients in Africa also have disseminated tuberculosis (infection throughout multiple organs). This type of tuberculosis is a significant cause of mortality in these patients. The purpose of this study is to evaluate the safety and effectiveness of a vaccine designed to prevent disseminated tuberculosis.

DETAILED DESCRIPTION:
Disseminated infection with Mycobacterium tuberculosis (dMTB) has been documented in 10% to 25% of patients with HIV infection in Africa. Unlike pulmonary tuberculosis (pMTB), most cases of dMTB are not recognized and death ensues rapidly. Therefore, dMTB may be a more important cause of HIV-associated mortality than pMTB in developing countries. Mycobacterium vaccae (MV) is an investigational vaccine prepared by heat inactivation of a nontuberculous mycobacteria. MV immunization may reduce the risk of HIV-associated dMTB. The purpose of this study is to define risk factors for HIV-associated dMTB and to assess the safety and effectiveness of an MV vaccine for the prevention of HIV-associated pulmonary and disseminated tuberculosis.

HIV positive patients with prior BCG immunization and HIV negative controls will be entered in a 5-year study in Tanzania. Participants will be randomized to receive a 5-dose series of MV or placebo over 12 months, with a repeat skin test at Month 14. Baseline evaluation will include medical history, chest x-ray, skin tests with purified protein derivative (PPD), and blood tests to evaluate interferon-gamma production. Participants with PPD reactions greater than or equal to 5 mm will receive 6 months of prophylaxis with isoniazid. Participants will be followed every 3 months for 3 to 5 years to assess new pMTB (microbiologic or clinical diagnosis) or dMTB (microbiologic diagnosis). Potential risk factors for dMTB will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* CD4 count more than 200 cells/mm3
* BCG scar

Exclusion Criteria:

* Active tuberculosis. Patients will be deferred from study enrollment until they show no signs of active disease.
* Serious underlying disease (e.g., congestive heart failure, advanced cancer)
* Life expectancy of less than 2 years
* Pregnancy. Women who are pregnant may be eligible for the study after they give birth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1975 (Actual)
Dates: Start 2001-09; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
safety and efficacy of a prime-boost immunization strategy for the prevention of HIV-associated dTB and pTB | every six months

SECONDARY OUTCOMES:
Risk factors for HIV-associated dTB and relative contributions of primary infection, reinfection, and reactivation in its pathogenesis | every six months

CONTACTS AND LOCATIONS:
Overall Officials: C. Fordham F von Reyn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Muhimbili University College of Health Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Result] Mtei L, Matee M, Herfort O, Bakari M, Horsburgh CR, Waddell R, Cole BF, Vuola JM, Tvaroha S, Kreiswirth B, Pallangyo K, von Reyn CF. High rates of clinical and subclinical tuberculosis among HIV-infected ambulatory subjects in Tanzania. Clin Infect Dis. 2005 May 15;40(10):1500-7. doi: 10.1086/429825. Epub 2005 Apr 12. PMID 15844073
- [Result] von Reyn CF, Mtei L, Arbeit RD, Waddell R, Cole B, Mackenzie T, Matee M, Bakari M, Tvaroha S, Adams LV, Horsburgh CR, Pallangyo K; DarDar Study Group. Prevention of tuberculosis in Bacille Calmette-Guerin-primed, HIV-infected adults boosted with an inactivated whole-cell mycobacterial vaccine. AIDS. 2010 Mar 13;24(5):675-85. doi: 10.1097/QAD.0b013e3283350f1b. PMID 20118767
- [Result] Lahey T, Arbeit RD, Bakari M, Horsburgh CR, Matee M, Waddell R, Mtei L, Vuola JM, Pallangyo K, von Reyn CF. Immunogenicity of a protective whole cell mycobacterial vaccine in HIV-infected adults: a phase III study in Tanzania. Vaccine. 2010 Nov 10;28(48):7652-8. doi: 10.1016/j.vaccine.2010.09.041. Epub 2010 Sep 25. PMID 20875492
- [Derived] Lahey T, Czechura T, Crabtree S, Arbeit RD, Matee M, Horsburgh CR, MacKenzie T, Bakari M, Pallangyo K, von Reyn CF. Greater preexisting interferon gamma responses to mycobacterial antigens and lower bacillary load during HIV-associated tuberculosis. J Infect Dis. 2013 Nov 15;208(10):1629-33. doi: 10.1093/infdis/jit396. Epub 2013 Aug 1. PMID 23908490
- [Derived] Lahey T, Mackenzie T, Arbeit RD, Bakari M, Mtei L, Matee M, Maro I, Horsburgh CR, Pallangyo K, von Reyn CF. Recurrent tuberculosis risk among HIV-infected adults in Tanzania with prior active tuberculosis. Clin Infect Dis. 2013 Jan;56(1):151-8. doi: 10.1093/cid/cis798. Epub 2012 Sep 12. PMID 22972862
- [Derived] Lahey T, Mitchell BK, Arbeit RD, Sheth S, Matee M, Horsburgh CR, MacKenzie T, Mtei L, Bakari M, Vuola JM, Pallangyo K, von Reyn CF. Polyantigenic interferon-gamma responses are associated with protection from TB among HIV-infected adults with childhood BCG immunization. PLoS One. 2011;6(7):e22074. doi: 10.1371/journal.pone.0022074. Epub 2011 Jul 20. PMID 21799772
- [Derived] von Reyn CF, Kimambo S, Mtei L, Arbeit RD, Maro I, Bakari M, Matee M, Lahey T, Adams LV, Black W, Mackenzie T, Lyimo J, Tvaroha S, Waddell R, Kreiswirth B, Horsburgh CR, Pallangyo K. Disseminated tuberculosis in human immunodeficiency virus infection: ineffective immunity, polyclonal disease and high mortality. Int J Tuberc Lung Dis. 2011 Aug;15(8):1087-92. doi: 10.5588/ijtld.10.0517. PMID 21740673
- [Derived] Lahey T, Sheth S, Matee M, Arbeit R, Horsburgh CR, Mtei L, Mackenzie T, Bakari M, Vuola JM, Pallangyo K, von Reyn CF. Interferon gamma responses to mycobacterial antigens protect against subsequent HIV-associated tuberculosis. J Infect Dis. 2010 Oct 15;202(8):1265-72. doi: 10.1086/656332. PMID 20812851
- [Derived] Lahey T, Matee M, Mtei L, Bakari M, Pallangyo K, von Reyn CF. Lymphocyte proliferation to mycobacterial antigens is detectable across a spectrum of HIV-associated tuberculosis. BMC Infect Dis. 2009 Feb 23;9:21. doi: 10.1186/1471-2334-9-21. PMID 19236695
- [Derived] Munseri PJ, Talbot EA, Mtei L, Fordham von Reyn C. Completion of isoniazid preventive therapy among HIV-infected patients in Tanzania. Int J Tuberc Lung Dis. 2008 Sep;12(9):1037-41. PMID 18713501